CLINICAL TRIAL: NCT00937170
Title: A Prospective, Randomized, Control Trial Comparing Total Knee Arthroplasty With Traditional and Gender-Specific Designs
Brief Title: Study Comparing Traditional and Gender-specific Total Knee Replacement Designs
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: Stryker Orthopaedics (Industry)
Responsible Party: R. Michael Meneghini, M.D., University of Connecticut Health Center Department of Orthopaedics
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09-036C-2; RMM001
Record Dates: First submitted 2009-07-09; First posted 2009-07-10 (Estimated); Last update posted 2011-01-21 (Estimated); Status verified 2011-01

CONDITIONS: Knee Osteoarthritis
Keywords: Total Knee Replacement; Gender Specific Design
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Gender Specific LPS flex (Experimental): Participants in this arm will receive the Zimmer LPS flex Gender Specific Implant design
  Interventions: Device: Zimmer LPS flex Gender Specific Implant (Total knee replacement)
- LPS flex (Active Comparator): Participants in this arm will receive the Zimmer High Flex LPS implant
  Interventions: Device: Zimmer High Flex LPS Implant (Total knee replacement)
- Triathlon (Active Comparator): Participants in this arm will receive the Stryker Triathlon Implant design
  Interventions: Device: Stryker Triathlon Implant (Total knee replacement)

INTERVENTIONS:
Device: Zimmer LPS flex Gender Specific Implant (Total knee replacement) — Outcomes comparison between a gender specific total knee implant, a standard total knee implant by the same company, and a standard total knee implant from another company
  Arms: Gender Specific LPS flex
Device: Zimmer High Flex LPS Implant (Total knee replacement) — Outcomes comparison between a gender specific total knee implant, a standard total knee implant by the same company, and a standard total knee implant from another company
  Arms: LPS flex
Device: Stryker Triathlon Implant (Total knee replacement) — Outcomes comparison between a gender specific total knee implant, a standard total knee implant by the same company, and a standard total knee implant from another company
  Arms: Triathlon

SUMMARY:
The purpose of this study is to compare results obtained with gender-specific and traditional knee replacement systems design among women undergoing total knee replacement surgery. Women who qualify and agree to participate will be randomly assigned to receive either a traditional or gender-specific knee replacement. During surgery, measurements of bone resection and bone-to-implant relationships will be recorded. At selected time intervals, participants will be asked to fill out questionnaires regarding pain and function, will be examined by their surgeon and routinely obtained xrays will be evaluated. In addition, a subset of participants will be randomly selected to undergo gait analysis to evaluate knee motion and muscle function.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of end-stage degenerative joint disease of the knee
* must be deemed appropriate for total knee replacement surgery

Exclusion Criteria:

* severe flexion deformity of the knee
* greater than 20deg varus or valgus malalignment
* osteomyelitis, septicemia, prior infection of the knee joint
* presence of infections or highly communicable diseases
* significant neurological or musculoskeletal disorders that affect gait or ability to bear weight on lower extremity
* metastatic disease
* congenital, developmental, bone disease or previous knee surgery that may interfere with the total knee prosthesis survival or success
* previous total knee replacement in affected knee
* arthrodesis of the affected knee

Ages: 40 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-06; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Evidence of improved pain relief and function | Pre-op, 4 weeks, 4 months, 1 year, 2 years

SECONDARY OUTCOMES:
Evidence of improved patellofemoral biomechanics | Pre-op, 4 months, 1 year

CONTACTS AND LOCATIONS:
Overall Officials: R. Michael Meneghini, M.D., Principal Investigator — University of Connecticut Health Center, Farmington CT, United States